CLINICAL TRIAL: NCT00071669
Title: Adjunctive Acupuncture as a Treatment for Bipolar Depression
Brief Title: Acupuncture as a Supplemental Treatment for Bipolar Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R03MH061589 (NIH); R03MH061589 (NIH); DSIR AT-SO
Record Dates: First submitted 2003-10-29; First posted 2003-10-30 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2005-11

CONDITIONS: Bipolar Disorder
Keywords: Mood Disorder; Acupuncture
MeSH Terms: conditions — Bipolar Disorder; Mood Disorders | interventions — Acupuncture Therapy

INTERVENTIONS:
Procedure: Acupuncture

SUMMARY:
The purpose of this study is to evaluate the effectiveness of acupuncture in the treatment of Bipolar Depression.

DETAILED DESCRIPTION:
Patients receive 8 weeks (12 sessions) of acupuncture treatment plus stable medication. Patients are randomly assigned to receive either acupuncture designed to relieve symptoms of depression or acupuncture designed to relieve some other legitimate physical condition. A comparison group of patients who take medication but do not receive acupuncture is assessed to evaluate the effectiveness of medication alone. Patients participate in clinical assessment each week, which includes visiting with a psychiatrist and completing symptom rating scales.

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM-IV criteria for bipolar I disorder or bipolar II disorder
* Demonstrate symptoms of depression as determined by a minimum score of 25 on the Inventory for Depressive Symptoms-Clinician Rated Scale
* Have taken stable psychoactive medications for at least 30 days prior to study entry

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30
Dates: Start 2001-11

CONTACTS AND LOCATIONS:
Locations (1):
- Bipolar Disorder Clinic and Research Program, Dallas, Texas, United States

REFERENCES:
- [Derived] Dennehy EB, Schnyer R, Bernstein IH, Gonzalez R, Shivakumar G, Kelly DI, Snow DE, Sureddi S, Suppes T. The safety, acceptability, and effectiveness of acupuncture as an adjunctive treatment for acute symptoms in bipolar disorder. J Clin Psychiatry. 2009 Jun;70(6):897-905. doi: 10.4088/JCP.08m04208. Epub 2009 May 5. PMID 19422756